CLINICAL TRIAL: NCT01493934
Title: Development of a Fast Measurement Technique of Insulin Resistance in Human, With 123-6-deoxy-6 Iodo-D-glucose, a New Tracer of Glucose Transport
Brief Title: Development of a Fast Measurement Technique of Insulin Resistance in Human
Acronym: GLUCIMAG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C09-07; 2009-014658-14 (EudraCT Number)
Record Dates: First submitted 2010-04-28; First posted 2011-12-16 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: metabolic syndrome; type 2 diabetes mellitus; insulin resistance; Scintigraphy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy volunteers (Active Comparator): First injection in human, on 6 healthy volunteers, sequentially : volunteer number1, then volunteers n°2 to n° 6, before infusion in type 2 diabetic patients.
  Interventions: Drug: injection of 6-DIG
- type 2 diabetic patients (Experimental): After completion of the study for the 6 healthy volunteers, infusion in 6 type 2 diabetic patients.
  Interventions: Drug: injection of 6-DIG

INTERVENTIONS:
Drug: injection of 6-DIG — Unique injection dose of 92.5 MBq

SUMMARY:
Insulin resistance, characterised by a depressed cellular sensitivity to insulin in insulin-sensitive organs, is a central feature of the metabolic syndrome. In people with no diabetes mellitus, the presence of metabolic syndrome leads to an increase of mortality, whatever the cause, but, as a majority, cardiovascular diseases.

In patients with type 2 diabetes mellitus, the presence of a metabolic syndrome leads to an increase in major adverse cardiovascular events. The prevalence of metabolic syndrome is led to grow in a near future, because of the increase of diabetes mellitus and obesity prevalence.

Actually, there is no simple tool to measure insulin resistance. The gold standard technique remains the hyperinsulinemic euglycemic clamp. However, the complexity and length of this technique render it unsuitable for routine clinical use. Many methods or index have been proposed to assess insulin resistance in human, but none have shown enough relevance to be used in clinical use.

Within the investigators U877 INSERM team, the investigators previously performed in vivo biodistribution studies with 6-DIG (6-deoxy-6-iodo-D-glucose), a new tracer of glucose transport, radiolabelled with123 iodine, with and without insulin, on the one hand in genetically diabetic mice (db/db), consequently having a severe insulin resistance and in the other hand in rats with acquired insulin resistance after a "fructose diet".

The investigators have demonstrated that 6-DIG is able to identify in vivo slight glucose transport variations in insulin sensible organs. Then, the investigators developed a fast and simple imaging protocol with a small animal gamma camera, which allows the obtaining of an insulin resistance index for each organ, directly transferable to human.

The investigators project is to transfer to human this measurement technique, perfectly validated in animal.

The main goal of this monocentric phase I-II study is to evaluate the tolerance to the insulin resistance measurement technique with 6DIG scintigraphy, in healthy volunteers and in diabetic patients. The investigators plan to enrol 6 healthy volunteers and 6 type 2 diabetic patients.

The investigators secondary goals will be to evaluate feasibility and reproducibility of the measurement technique, to follow pharmacokinetic and to assess efficacy of 6-DIG to measure insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged between 35 et 60 years old
* Body mass index between 20 and 25
* Waist measurement < 94 cm for men and < 80 cm for women
* Normal basal glycemia, between 3,8 and 5,8 mmol/l
* Normal basal insulinemia, between 3 and 13 μUI/ml
* HbA1c < 6%
* Total cholesterol < 2 g/l
* LDL cholesterol < 1,6 g/l
* HDL cholesterol 0,4 g/l for men and 0,5 g/l for women
* Triglyceride level < 1,5 g/l
* For women not menopausal since at last one year or not surgically sterilised:

On-going contraception, physical or hormonal, excepted local methods (spermicidal, diaphragm, condom, cape)

* Type 2 diabetic patients
* Aged between 35 et 60 years old
* Stable type 2 diabetes mellitus: no ketoacidosis sign during last month
* HbA1c between 6 and 8% during the 3 months before study inclusion
* Monotherapy by metformin or diet only
* For women not menopausal since at last one year or not surgically sterilised:
* On-going contraception, physical or hormonal, excepted local methods (spermicidal, diaphragm, condom, cape)

Exclusion Criteria:

* Diabetes mellitus previously known
* Other on-going progressive illness
* Psychiatric illness, needing a chronic treatment
* Previous history of myocardial infarction, coronary artery disease, cardiac rhythm troubles, stroke, epilepsy, cranial trauma, pituitary surgery, disease likely to reduce the ability of absorption, diffusion or excretion of the radiotracer.
* Severe hypertension defined by par SAP > 180 mmHg and/or DAP > 110 mmHg
* Allergy to one of the components of the products used during the study
* Nuclear medicine examination during the 30 days prior to study inclusion
* Treatment likely to interfere with glucose metabolism
* Alcohol or drug intoxication
* Vegetarian or restrictive low-calory diet,
* Pregnant, parturient or breast-feeding women,
* Inappropriate way of life
* Type 2 diabetic patients.
* Previous history of myocardial infarction
* Severe hypertension defined by par SAP > 180 mmHg and/or DAP > 110 mmHg
* Previous history of coronary artery disease, cardiac rhythm troubles, stroke, epilepsy, cranial trauma, pituitary surgery, disease likely to reduce the ability of absorption, diffusion or excretion of the radiotracer.
* Psychiatric illness, needing a chronic treatment
* On-going insulin treatment
* On-going treatment other than metformin, likely to interfere with glucose metabolism
* Previous history of disease likely to reduce the ability of absorption, diffusion or excretion of the radiotracer
* Allergy to one of the components of the products used during the study
* Nuclear medicine examination during the 30 days prior to study inclusion
* Alcohol or drug intoxication
* Vegetarian or restrictive low-calory diet,
* Pregnant, parturient or breast-feeding women,
* Inappropriate way of life

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change of glycemia | Before inclusion in clinical trial, Before radiotracer injection, After radiotracer injection (time: 30s, 1', 2',5',10',15',25', 1 hour, 2 hours, 4 hours, 8 hours, 24 hours)
  Assessment of tolerance to insulin resistance measurement technique with 6-DIG scintigraphy, in healthy volunteers
  * clinical tolerance to 6-DIG infusion
  * clinical and biological tolerance to insulin infusion
  * evaluation of dosimetry

SECONDARY OUTCOMES:
insulinemia | Before inclusion in clinical trial, Before radiotracer injection, After radiotracer injection (time: 30s, 1', 2',5',10',15',25', 1 hour, 2 hours, 4 hours, 8 hours, 24 hours)
clinical side effects | Before inclusion in clinical trial, Before radiotracer injection, After radiotracer injection (time: 30s, 1', 2',5',10',15',25', 1 hour, 2 hours, 4 hours, 8 hours, 24 hours)
  hypoglycemia symptoms
dosimetry | during the 24 hours following injection of 6-DIG
  organs biodistribution of radioactivity
insulin resistance | 0-15 minutes following 6-DIG infusion
  scintigraphic measurement of glucose transport in heart before and after infusion of insulin

CONTACTS AND LOCATIONS:
Overall Officials: Alex Calizzano, MD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Alex Calizzano, MD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Service de Biophysique et Médecine Nucléaire, CHU de Grenoble, Grenoble, France

REFERENCES:
- [Background] Calizzano A, Perret P, Desruet MD, Ahmadi M, Reboulet G, Djaileb L, Vanzetto G, Fagret D, Barone-Rochette G, Ghezzi C. Safety, Biodistribution, and Dosimetry of 123I-6-Deoxy-6-Iodo-D-Glucose, a Tracer of Glucose Transport, in Healthy and Diabetic Volunteers. Clin Nucl Med. 2019 May;44(5):386-393. doi: 10.1097/RLU.0000000000002510. PMID 30888989